CLINICAL TRIAL: NCT04888793
Title: Immune Response to Anti COVID-19 Vaccine in Immunocompromised Patients: a Cohort Study
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 210405014
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-05

CONDITIONS: Covid19; COVID-19 Vaccines
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cancer Patients on active treatment
  Interventions: Diagnostic Test: Serologic immune response evaluation
- Bone marrow transplant patients
  Interventions: Diagnostic Test: Serologic immune response evaluation
- Solid organ transplant recipients
  Interventions: Diagnostic Test: Serologic immune response evaluation
- HIV patients
  Interventions: Diagnostic Test: Serologic immune response evaluation
- Rheumatic disease patients
  Interventions: Diagnostic Test: Serologic immune response evaluation
- Healthy controls
  Interventions: Diagnostic Test: Serologic immune response evaluation

INTERVENTIONS:
Diagnostic Test: Serologic immune response evaluation — Detection of total and neutralizing antibodies against SARS-CoV-2

SUMMARY:
Despite COVID-19 pandemic having started more than one year ago, there are still limited treatment options for these patients, and over 145 million cases and 3 millions deaths have ensued worldwide. Fortunately, SARSCoV2 vaccines have been developed at an unprecedented pace. While the vaccination programs are still ongoing, early reports on efficacy are mainly centered on healthy population. In Chile most people have received the inactivated Coronavac vaccine. Data on the immune response after vaccination in immunocompromised patients is lacking. Therefore, this study aims to evaluate the immune response after Coronavac vaccine in 5 cohorts of immunocompromised patients and healthy controls. We will include patients with cancer, HIV, solid organ transplant and patients receiving immunomodulatory agents for rheumatic diseases.

ELIGIBILITY:
General Inclusion Criteria:

* Eastern Cooperative Oncology Group < 3
* Vaccination with 2 doses of Coronavac vaccine

General Exclusion Criteria:

* Previous SARS-CoV-2 infection
* Vaccination with Coronavac more than 12 weeks before informed consent
* Intravenous immunoglobulin therapy 60 days before informed consent
* Any condition, that could interfere with the participant's participation during the study in the opinion of the treating investigator.

Cancer Cohort

Inclusion Criteria:

* Diagnosis of cancer in the previous 5 years (consistent biopsy is required).
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Bone marrow transplant, solid organ recipient, HIV, immunosuppressant treatment for other condition.

Bone Marrow Transplant Cohort

Inclusion Criteria:

* Bone marrow transplant between January 2019 and December 2020

Exclusion Criteria:

* Other cancer diagnosis during the last 5 years, solid organ recipient, HIV, immunosuppressant treatment for other condition.

Solid Organ Recipient Cohort:

Inclusion Criteria:

* Liver, kidney or heart transplant between January 2019 and December 2020
* Active immunosuppressant treatment

Exclusion Criteria:

- Cancer diagnosis during the last 5 years, bone marrow transplant, immunosuppressant treatment for other condition, HIV

HIV Cohort:

Inclusion Criteria:

* CD4 <= 500 cels/mm3 documented one year before study enrollment
* Active antiretroviral therapy
* Viral load < 200 copies/ml

Exclusion Criteria:

* Cancer diagnosis during the last 5 years, bone marrow transplant or solid organ recipient, immunosuppressant treatment.

Rheumatic Disease Cohort

Inclusion Criteria:

* Diagnosis of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, relapsing polychondritis, Behcet disease or juvenile idiopathic arthritis
* Chronic immunomodulatory treatment with anti-TNF, anti-IL6 or anti-IL17 agents

Exclusion Criteria:

* Treatment with more than one biological agent.
* Cancer diagnosis during the last 5 years, bone marrow transplant or solid organ recipient, HIV diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at the Red de Salud UC Christus in Santiago, Chile will be invited.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of positive neutralizing antibodies 8 to12 weeks after Coronavac vaccine | 8 to12 weeks after Coronavac vaccine

SECONDARY OUTCOMES:
Neutralizing geometric mean titers 8 to12 weeks after Coronavac vaccine | 8 to12 weeks after Coronavac vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Balcells, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Red de Salud UC Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balcells ME, Le Corre N, Duran J, Ceballos ME, Vizcaya C, Mondaca S, Dib M, Rabagliati R, Sarmiento M, Burgos PI, Espinoza M, Ferres M, Martinez-Valdebenito C, Ruiz-Tagle C, Ortiz C, Ross P, Budnik S, Solari S, Vizcaya MLA, Lembach H, Berrios-Rojas R, Melo-Gonzalez F, Rios M, Kalergis AM, Bueno SM, Nervi B. Reduced Immune Response to Inactivated Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine in a Cohort of Immunocompromised Patients in Chile. Clin Infect Dis. 2022 Aug 24;75(1):e594-e602. doi: 10.1093/cid/ciac167. PMID 35255140